CLINICAL TRIAL: NCT04911712
Title: The Effectiveness of a High-Protein Liquid Dietary Supplementation in Improving Nutritional Status of Malnourished Patients in Hospital Care: a Preliminary Study
Brief Title: The Effectiveness of a High-Protein Liquid Dietary Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MARCELLUS SIMADIBRATA (Other)
Responsible Party: Sponsor-Investigator, MARCELLUS SIMADIBRATA, Prof. dr. Marcellus Simadibrata Ph.D, Sp.PD-KGEH, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KET-313/UN2.F1/ETIK
Record Dates: First submitted 2021-04-01; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Malnutrition; Nutritional Status; Hospital; Hand Strength; Body Mass Index; Nutrition Assessment
Keywords: Malnutrition; high-protein diet; nutritional status; hospitals; hand strength; body mass index; nutrition assessment; preliminary data
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: a Preliminary Study
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Randomly selected malnourished patients for normal protein liquid diet supplementation (Active Comparator): Randomly selected malnourished patients for normal protein liquid diet supplementation
  Interventions: Dietary Supplement: a hospital formula of normal protein liquid diet supplementation
- Randomly selected Malnourished patients with high protein liquid diet supplementation (Experimental): Malnourished patients with high protein liquid diet supplementation
  Interventions: Dietary Supplement: a hospital formula of high protein liquid food supplementation

INTERVENTIONS:
Dietary Supplement: a hospital formula of normal protein liquid diet supplementation — group 1 (control group) who will get a hospital formula of normal protein liquid diet supplementation (40 grams per 1000 mL)
  Arms: Randomly selected malnourished patients for normal protein liquid diet supplementation
Dietary Supplement: a hospital formula of high protein liquid food supplementation — group 2 (intervention group) will get a hospital formula of high protein liquid food supplementation (60 grams per 1000 mL) as much as 2 bottles (each bottle contains 200 mL)
  Arms: Randomly selected Malnourished patients with high protein liquid diet supplementation

SUMMARY:
This study was a double-blind randomized controlled trial conducted to assess the effectiveness of high protein liquid dietary supplementation in malnourished hospitalized patients. The patients were assessed for their nutritional status based on ESPEN 2015 criteria. Patients who experienced malnutrition will be divided into 2 groups, namely the control group which was given a normal protein liquid diet, while the intervention group was given high protein liquid diet supplementation as much as 2 bottles (200 mL) per day for 7-10 days. Furthermore, the nutritional status of the patient was assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 18 years old to 60 years old
2. Malnutrition hospitalized patient based on European Society for Clinical Nutrition and Metabolism (ESPEN) 2015 criteria
3. Agreed to participate

Exclusion Criteria:

1. Malignancy
2. Chronic kidney disease stage III-V
3. Decompensated hepatic cirrhosis
4. Allergic to milk or lactose intolerance
5. Could not be randomised and participate in this study by clinical judgement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Right handgrip strength | Handgrip strength is assessed at day 10 of dietary administration supplementation in each arm
  Handgrip strength in kg based on sex and age
Adult malnutrition classification according to the WHO | the classification of malnutrition is assessed at day 10 of dietary supplementation in each arm
  The classification of Adult malnutrition according to the WHO based on BMI which categorized into (mild,moderate or severe)
Nutritional status based on Subjective Global Assessment (SGA) | All SGA assesment is done at day 10 of dietary supplementation in each arm
  the Nutritional status based on Subjective Global Assessment (SGA). Group A is classified as Normal/ well-nourished. Group B is classified as Mild-Moderate nutrition. Group C is classified as Severe malnutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meijers JM, van Bokhorst-de van der Schueren MA, Schols JM, Soeters PB, Halfens RJ. Defining malnutrition: mission or mission impossible? Nutrition. 2010 Apr;26(4):432-40. doi: 10.1016/j.nut.2009.06.012. Epub 2009 Dec 1. PMID 19954929
- [Background] Allard JP, Keller H, Jeejeebhoy KN, Laporte M, Duerksen DR, Gramlich L, Payette H, Bernier P, Vesnaver E, Davidson B, Teterina A, Lou W. Malnutrition at Hospital Admission-Contributors and Effect on Length of Stay: A Prospective Cohort Study From the Canadian Malnutrition Task Force. JPEN J Parenter Enteral Nutr. 2016 May;40(4):487-97. doi: 10.1177/0148607114567902. Epub 2015 Jan 26. PMID 25623481
- [Background] Alvarez-Hernandez J, Planas Vila M, Leon-Sanz M, Garcia de Lorenzo A, Celaya-Perez S, Garcia-Lorda P, Araujo K, Sarto Guerri B; PREDyCES researchers. Prevalence and costs of malnutrition in hospitalized patients; the PREDyCES Study. Nutr Hosp. 2012 Jul-Aug;27(4):1049-59. doi: 10.3305/nh.2012.27.4.5986. PMID 23165541
- [Background] Schindler K, Pernicka E, Laviano A, Howard P, Schutz T, Bauer P, Grecu I, Jonkers C, Kondrup J, Ljungqvist O, Mouhieddine M, Pichard C, Singer P, Schneider S, Schuh C, Hiesmayr M; NutritionDay Audit Team. How nutritional risk is assessed and managed in European hospitals: a survey of 21,007 patients findings from the 2007-2008 cross-sectional nutritionDay survey. Clin Nutr. 2010 Oct;29(5):552-9. doi: 10.1016/j.clnu.2010.04.001. PMID 20434820
- [Background] Lim SL, Ong KC, Chan YH, Loke WC, Ferguson M, Daniels L. Malnutrition and its impact on cost of hospitalization, length of stay, readmission and 3-year mortality. Clin Nutr. 2012 Jun;31(3):345-50. doi: 10.1016/j.clnu.2011.11.001. Epub 2011 Nov 26. PMID 22122869
- [Background] Garber AK, Mauldin K, Michihata N, Buckelew SM, Shafer MA, Moscicki AB. Higher calorie diets increase rate of weight gain and shorten hospital stay in hospitalized adolescents with anorexia nervosa. J Adolesc Health. 2013 Nov;53(5):579-84. doi: 10.1016/j.jadohealth.2013.07.014. Epub 2013 Sep 17. PMID 24054812
- [Background] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Background] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486
- [Background] Detsky AS, McLaughlin JR, Baker JP, Johnston N, Whittaker S, Mendelson RA, Jeejeebhoy KN. What is subjective global assessment of nutritional status? JPEN J Parenter Enteral Nutr. 1987 Jan-Feb;11(1):8-13. doi: 10.1177/014860718701100108. PMID 3820522
- [Background] Huynh DT, Devitt AA, Paule CL, Reddy BR, Marathe P, Hegazi RA, Rosales FJ. Effects of oral nutritional supplementation in the management of malnutrition in hospital and post-hospital discharged patients in India: a randomised, open-label, controlled trial. J Hum Nutr Diet. 2015 Aug;28(4):331-43. doi: 10.1111/jhn.12241. Epub 2014 May 9. PMID 24809429